CLINICAL TRIAL: NCT05910515
Title: Improving Performance in Pediatric Trauma by Teaching Nontechnical Skills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dan Poenaru, Principal investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-7561
Record Dates: First submitted 2023-05-23; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Injuries
Keywords: child; non-technical skills; pediatric trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Regular debriefing
- Intervention (Experimental): Structured debriefing in non-technical skills
  Interventions: Other: Debriefing

INTERVENTIONS:
Other: Debriefing — Structured debriefing in non-technical skills. (This is an educational study)
  Arms: Intervention

SUMMARY:
The goal of this trial is to test a debriefing protocol to improve non-technical skills (NTS) in medical students. The study aims to answer the following questions:

* Does a debriefing intervention improve medical students' NTS?
* Does the intervention have an impact on the students' performance in simulated scenarios?

Participants in the study will be randomly assigned to one of the teams, each consisting of a trauma team leader and three assistants. The teams will rotate across four different scenarios, allowing participants to switch roles and act as team leaders. The intervention teams will be debriefed using the study protocol, while the control groups will receive standard technical feedback without focusing on NTS.

The primary outcome measure will be the Non-Technical Skills for Surgeons (NOTSS) score, which is a validated assessment tool for NTS. Secondary outcome measures include the number of correct interventions performed in each scenario.

The study will involve 40 medical students, and the sample size was determined based on previous studies and statistical considerations. A panel of health educators will define the debriefing protocol, and the trial has been approved by the McGill Research Ethics Board office.

The study findings are expected to contribute significantly to the training of providers of trauma care for children worldwide. By exploring the impact of debriefing on NTS in pediatric trauma education, this project aims to fill a critical gap in current training models.

DETAILED DESCRIPTION:
BACKGROUND AND STUDY RATIONALE Pediatric trauma is a global epidemic, and improving pediatric trauma care requires a focus on healthcare provider education. Studies have shown that inadequate training and poor non-technical skills contribute to errors in trauma care. Non-technical skills, including teamwork communication, leadership, situational awareness, and decision-making, are crucial in delivering effective healthcare.

These skills were initially recognized in the aviation industry and have since been studied and applied in various settings. However, the intentional teaching of non-technical skills in healthcare contexts is lacking. While medical content and technical skills have transitioned from the classroom to practical settings and simulation labs, non-technical skills have not received the same attention, leading to suboptimal quality of medical care.

The Non-Technical Skills for Surgeons (NOTSS) is a valuable tool for assessing these skills in surgeons. It employs a numeric scale to score surgeons' attitudes, enabling educators to identify strengths and weaknesses. NOTSS evaluates four main behavioral categories: situation awareness, decision-making, teamwork, and leadership. Each category consists of four elements that are assessed based on the original NOTSS handbook. Adequate performance is indicated by a score above 0.7 in each category. This scoring system facilitates personalized feedback and highlights areas for improvement.

Although NOTSS is primarily used in the operating room rather than in simulation training, there is currently a lack of studies evaluating the training of non-technical skills in pediatric trauma courses. This highlights the need to develop educational resources specifically focused on teaching non-technical skills in pediatric trauma education.

OBJECTIVES & HYPOTHESIS

The hypothesis of this study is that teaching and evaluating non-technical skills in pediatric trauma scenarios will enhance the overall clinical performance of medical students and general surgery trainees. The study aims to achieve the following objectives:

1. Assess the ratings of medical students and general surgery trainees using the Non-Technical Skills for Surgeons (NOTSS) assessment tool.
2. Investigate the impact of individual differences, such as training experience, on NOTSS scores.
3. Evaluate the effectiveness of standardized debriefing sessions in improving NOTSS scores and outcomes in simulated assessments of pediatric trauma.

STUDY METHODS

Study Design:

The study will be a randomized controlled trial using the NOTSS score and debriefing strategies. Two rounds of pediatric trauma-simulated scenarios will be conducted. After the first round, participants will be randomly assigned to either an intervention group or a control group. The intervention group will receive formal debriefing on non-technical and technical performance, while the control group will only receive feedback on technical skills.

Participant Recruitment:

Collaboration will be sought from the McGill Faculty of Medicine and Health Sciences Undergraduate Education Office and the McGill Postgraduate Education Office to invite students and residents to participate. Flyers will be displayed, and announcements will be made on social media. In Brazil, invitations will be sent via email lists of participating universities and social media platforms.

Study Duration:

The study is expected to run from September 1, 2022, to September 1, 2024.

Data Analysis:

Data will be collected using Microsoft Forms, Excel, and Word, and analyzed using R version 3.2.5. Descriptive analysis will be conducted for participants' profile features and outcome variables. Inferential analysis will compare data before and after intervention/debriefings, between medical students and surgical residents, and between control and intervention groups using appropriate statistical tests.

Ethical Considerations:

The study will adhere to ethical guidelines and receive approval from the relevant ethics boards. Confidentiality measures will be implemented, and informed consent will be obtained from all participants. Data will be deidentified, stored securely, and destroyed after the study's completion. A dissemination plan is in place, targeting the academic community, policymakers, and the general public, while ensuring participant anonymity.

ELIGIBILITY:
Inclusion Criteria:

1. Canadian cohort

   * McGill University, years 3 or 4 medical students. or
   * McGill University Health Centre general surgery residents
2. Brazilian cohort

   * Medical students, years 5 or 6. or
   * Brazilian general surgery residents

Exclusion Criteria:

1. Canadian cohort

   * Medical students of years 1 and 2;
   * Residents that are not from the General Surgery service;
2. Brazilian cohort

   * Medical students of years 1, 2, 3 & 4.
   * Residents that are not from the General Surgery service;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, female, non-binary
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
NOTSS score | During the student's participation in the simulated scenarios (four hours)
  The Non-technical skills for surgeons (NOTSS) score evaluates four major categories of non-technical skills: situation awareness, decision-making, teamwork, and leadership. Each category is assessed based on specific elements outlined in the NOTSS handbook (www.notss.org). It is a continuous variable ranging from 1 to 4. Higher scores on the NOTSS scale indicate better non-technical skills, while lower scores suggest areas that may need improvement. Educators are responsible for observing the trainees and scoring their behaviors during the simulated scenarios.

SECONDARY OUTCOMES:
Number of interventions performed | During the student's participation in the simulated scenarios (four hours)
  The evaluation of student performance in each simulated scenario involves a total of 12 steps. The number of steps successfully completed by the student will be recorded and expressed as a percentage for each scenario. This measurement provides an objective assessment of the student's ability to effectively carry out the required tasks in the given scenario.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Poenaru, Principal Investigator — McGill
Locations (2):
- Medical schools in Brazil, Belo Horizonte, Brazil
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Once study is published, according to the journal's/editor's policies.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Global Burden of Disease Child and Adolescent Health Collaboration; Kassebaum N, Kyu HH, Zoeckler L, Olsen HE, Thomas K, Pinho C, Bhutta ZA, Dandona L, Ferrari A, Ghiwot TT, Hay SI, Kinfu Y, Liang X, Lopez A, Malta DC, Mokdad AH, Naghavi M, Patton GC, Salomon J, Sartorius B, Topor-Madry R, Vollset SE, Werdecker A, Whiteford HA, Abate KH, Abbas K, Damtew SA, Ahmed MB, Akseer N, Al-Raddadi R, Alemayohu MA, Altirkawi K, Abajobir AA, Amare AT, Antonio CAT, Arnlov J, Artaman A, Asayesh H, Avokpaho EFGA, Awasthi A, Ayala Quintanilla BP, Bacha U, Betsu BD, Barac A, Barnighausen TW, Baye E, Bedi N, Bensenor IM, Berhane A, Bernabe E, Bernal OA, Beyene AS, Biadgilign S, Bikbov B, Boyce CA, Brazinova A, Hailu GB, Carter A, Castaneda-Orjuela CA, Catala-Lopez F, Charlson FJ, Chitheer AA, Choi JJ, Ciobanu LG, Crump J, Dandona R, Dellavalle RP, Deribew A, deVeber G, Dicker D, Ding EL, Dubey M, Endries AY, Erskine HE, Faraon EJA, Faro A, Farzadfar F, Fernandes JC, Fijabi DO, Fitzmaurice C, Fleming TD, Flor LS, Foreman KJ, Franklin RC, Fraser MS, Frostad JJ, Fullman N, Gebregergs GB, Gebru AA, Geleijnse JM, Gibney KB, Gidey Yihdego M, Ginawi IAM, Gishu MD, Gizachew TA, Glaser E, Gold AL, Goldberg E, Gona P, Goto A, Gugnani HC, Jiang G, Gupta R, Tesfay FH, Hankey GJ, Havmoeller R, Hijar M, Horino M, Hosgood HD, Hu G, Jacobsen KH, Jakovljevic MB, Jayaraman SP, Jha V, Jibat T, Johnson CO, Jonas J, Kasaeian A, Kawakami N, Keiyoro PN, Khalil I, Khang YH, Khubchandani J, Ahmad Kiadaliri AA, Kieling C, Kim D, Kissoon N, Knibbs LD, Koyanagi A, Krohn KJ, Kuate Defo B, Kucuk Bicer B, Kulikoff R, Kumar GA, Lal DK, Lam HY, Larson HJ, Larsson A, Laryea DO, Leung J, Lim SS, Lo LT, Lo WD, Looker KJ, Lotufo PA, Magdy Abd El Razek H, Malekzadeh R, Markos Shifti D, Mazidi M, Meaney PA, Meles KG, Memiah P, Mendoza W, Abera Mengistie M, Mengistu GW, Mensah GA, Miller TR, Mock C, Mohammadi A, Mohammed S, Monasta L, Mueller U, Nagata C, Naheed A, Nguyen G, Nguyen QL, Nsoesie E, Oh IH, Okoro A, Olusanya JO, Olusanya BO, Ortiz A, Paudel D, Pereira DM, Perico N, Petzold M, Phillips MR, Polanczyk GV, Pourmalek F, Qorbani M, Rafay A, Rahimi-Movaghar V, Rahman M, Rai RK, Ram U, Rankin Z, Remuzzi G, Renzaho AMN, Roba HS, Rojas-Rueda D, Ronfani L, Sagar R, Sanabria JR, Kedir Mohammed MS, Santos IS, Satpathy M, Sawhney M, Schottker B, Schwebel DC, Scott JG, Sepanlou SG, Shaheen A, Shaikh MA, She J, Shiri R, Shiue I, Sigfusdottir ID, Singh J, Silpakit N, Smith A, Sreeramareddy C, Stanaway JD, Stein DJ, Steiner C, Sufiyan MB, Swaminathan S, Tabares-Seisdedos R, Tabb KM, Tadese F, Tavakkoli M, Taye B, Teeple S, Tegegne TK, Temam Shifa G, Terkawi AS, Thomas B, Thomson AJ, Tobe-Gai R, Tonelli M, Tran BX, Troeger C, Ukwaja KN, Uthman O, Vasankari T, Venketasubramanian N, Vlassov VV, Weiderpass E, Weintraub R, Gebrehiwot SW, Westerman R, Williams HC, Wolfe CDA, Woodbrook R, Yano Y, Yonemoto N, Yoon SJ, Younis MZ, Yu C, Zaki MES, Zegeye EA, Zuhlke LJ, Murray CJL, Vos T. Child and Adolescent Health From 1990 to 2015: Findings From the Global Burden of Diseases, Injuries, and Risk Factors 2015 Study. JAMA Pediatr. 2017 Jun 1;171(6):573-592. doi: 10.1001/jamapediatrics.2017.0250. PMID 28384795
- [Background] Kiragu AW, Dunlop SJ, Wachira BW, Saruni SI, Mwachiro M, Slusher T. Pediatric Trauma Care in Low- and Middle-Income Countries: A Brief Review of the Current State and Recommendations for Management and a Way Forward. J Pediatr Intensive Care. 2017 Mar;6(1):52-59. doi: 10.1055/s-0036-1584676. Epub 2016 Jun 24. PMID 31073425
- [Background] Kiragu AW, Dunlop SJ, Mwarumba N, Gidado S, Adesina A, Mwachiro M, Gbadero DA, Slusher TM. Pediatric Trauma Care in Low Resource Settings: Challenges, Opportunities, and Solutions. Front Pediatr. 2018 Jun 4;6:155. doi: 10.3389/fped.2018.00155. eCollection 2018. PMID 29915778
- [Background] Roberts NK, Williams RG, Schwind CJ, Sutyak JA, McDowell C, Griffen D, Wall J, Sanfey H, Chestnut A, Meier AH, Wohltmann C, Clark TR, Wetter N. The impact of brief team communication, leadership and team behavior training on ad hoc team performance in trauma care settings. Am J Surg. 2014 Feb;207(2):170-8. doi: 10.1016/j.amjsurg.2013.06.016. Epub 2013 Oct 2. PMID 24468024
- [Background] Ziesmann MT, Widder S, Park J, Kortbeek JB, Brindley P, Hameed M, Paton-Gay JD, Engels PT, Hicks C, Fata P, Ball CG, Gillman LM. S.T.A.R.T.T.: development of a national, multidisciplinary trauma crisis resource management curriculum-results from the pilot course. J Trauma Acute Care Surg. 2013 Nov;75(5):753-8. doi: 10.1097/TA.0b013e3182a925df. PMID 24158191
- [Background] Higashi H, Barendregt JJ, Kassebaum NJ, Weiser TG, Bickler SW, Vos T. Burden of injuries avertable by a basic surgical package in low- and middle-income regions: a systematic analysis from the Global Burden of Disease 2010 Study. World J Surg. 2015 Jan;39(1):1-9. doi: 10.1007/s00268-014-2685-x. PMID 25008243
- [Background] Lee A, Finstad A, Gawad N, Boet S, Raiche I, Balaa F. Nontechnical Skills (NTS) in the Undergraduate Surgical and Anesthesiology Curricula: Are We Adequately Preparing Medical Students? J Surg Educ. 2021 Mar-Apr;78(2):502-511. doi: 10.1016/j.jsurg.2020.08.001. Epub 2020 Aug 21. PMID 32839149
- [Background] Jung JJ, Borkhoff CM, Juni P, Grantcharov TP. Non-Technical Skills for Surgeons (NOTSS): Critical appraisal of its measurement properties. Am J Surg. 2018 Nov;216(5):990-997. doi: 10.1016/j.amjsurg.2018.02.021. Epub 2018 Feb 17. PMID 29478826
- [Background] Patel EA, Aydin A, Desai A, Dasgupta P, Ahmed K. Current status of simulation-based training in pediatric surgery: A systematic review. J Pediatr Surg. 2019 Sep;54(9):1884-1893. doi: 10.1016/j.jpedsurg.2018.11.019. Epub 2018 Dec 8. PMID 30573294
- [Background] Helmreich RL, Merritt AC, Wilhelm JA. The evolution of Crew Resource Management training in commercial aviation. Int J Aviat Psychol. 1999;9(1):19-32. doi: 10.1207/s15327108ijap0901_2. PMID 11541445
- [Background] Sevdalis N, Davis R, Koutantji M, Undre S, Darzi A, Vincent CA. Reliability of a revised NOTECHS scale for use in surgical teams. Am J Surg. 2008 Aug;196(2):184-90. doi: 10.1016/j.amjsurg.2007.08.070. Epub 2008 Jun 16. PMID 18558392
- [Background] Jensen AR, McLaughlin C, Subacius H, McAuliff K, Nathens AB, Wong C, Meeker D, Burd RS, Ford HR, Upperman JS. Simulation-based training is associated with lower risk-adjusted mortality in ACS pediatric TQIP centers. J Trauma Acute Care Surg. 2019 Oct;87(4):841-848. doi: 10.1097/TA.0000000000002433. PMID 31589193
- [Background] Yule S, Paterson-Brown S. Surgeons' non-technical skills. Surg Clin North Am. 2012 Feb;92(1):37-50. doi: 10.1016/j.suc.2011.11.004. Epub 2011 Dec 28. PMID 22269259
- [Background] Leenstra NF, Jung OC, Cnossen F, Jaarsma ADC, Tulleken JE. Development and Evaluation of the Taxonomy of Trauma Leadership Skills-Shortened for Observation and Reflection in Training: A Practical Tool for Observing and Reflecting on Trauma Leadership Performance. Simul Healthc. 2021 Feb 1;16(1):37-45. doi: 10.1097/SIH.0000000000000474. PMID 32732816
- [Background] Sanfey H. Assessment of surgical training. Surgeon. 2014 Dec;12(6):350-6. doi: 10.1016/j.surge.2014.07.001. Epub 2014 Jul 31. PMID 25087505